CLINICAL TRIAL: NCT05617872
Title: Vinegar-induced Collection of Duodenal Pancreatic Juice Via Endoscopic Ultrasound
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wu Xi, Associated Professor, M.D., Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: K2379
Record Dates: First submitted 2022-11-06; First posted 2022-11-16 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; Endoscopic ultrasound; pancreatic juice
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Acetic Acid; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Normal Saline Group (Placebo Comparator): Inject 20ml normal saline solution into duodenum and collect the pancreatic juice for 15 minutes via EUS, changing the collection bottle every 5 minutes.
  Interventions: Drug: Saline (NaCl 0,9 %) (placebo)
- Vinegar 20ml Group (Experimental): Inject 20ml vinegar (5% acetic acid solution) into duodenum and collect the pancreatic juice for 15 minutes via EUS, changing the collection bottle every 5 minutes.
  Interventions: Drug: Vinegar 20ml
- Vinegar 40ml Group (Active Comparator): Inject 40ml vinegar (5% acetic acid solution) into duodenum and collect the pancreatic juice for 15 minutes via EUS, changing the collection bottle every 5 minutes.
  Interventions: Drug: Vinegar 40ml

INTERVENTIONS:
Drug: Vinegar 20ml — Inject 20ml vinegar (5% acetic acid solution) into duodenum and collect the pancreatic juice for 15 minutes via EUS, changing the collection bottle every 5 minutes.
  Arms: Vinegar 20ml Group
Drug: Saline (NaCl 0,9 %) (placebo) — Inject 20ml normal saline solution into duodenum and collect the pancreatic juice for 15 minutes via EUS, changing the collection bottle every 5 minutes.
  Arms: Normal Saline Group
Drug: Vinegar 40ml — Inject 40ml vinegar (5% acetic acid solution) into duodenum and collect the pancreatic juice for 15 minutes via EUS, changing the collection bottle every 5 minutes.
  Arms: Vinegar 40ml Group

SUMMARY:
The goal of this clinical trial is to learn about the feasibility of collecting pancreatic juice through duodenal aspiration by ultrasound endoscopy (EUS) for molecular marker testing after intraduodenal infusion of vinegar in patients with suspected pancreatic cancer and who are scheduled to have endoscopic ultrasound with fine needle aspiration (EUS-FNA). The main questions it aims to answer are:

* Is vinegar-induced collection of duodenal pancreatic juice via endoscopic ultrasound feasible?
* What is the best operating condition (amount of vinegar, collection time, etc.) of vinegar-induced collection of duodenal pancreatic juice via endoscopic ultrasound?

Participants will have EUS as scheduled, during which different amount of vinegar will be infused into duodenum and then pancreatic juice be collected for different time via suction by EUS.

Researchers will compare the amount of collected pancreatic juice and molecular marker level in different groups to determine the best operating condition for vinegar-induced collection of duodenal pancreatic juice via endoscopic ultrasound.

DETAILED DESCRIPTION:
This is a single center, prospective, randomized-controlled study. Participants who are diagnosed as suspected pancreatic cancer and are schedule to have EUS-FNA will have saline or different amount of vinegar infused into duodenum and pancreatic juiced collected via EUS suction during different period of time under intravenous anesthesia.

The collected pancreatic juice will be weighed instantly and frozen in 10 minutes under -80℃ for further tests.

Researchers will compare the weight, cfDNA (cell free DNA) concentration, PLA2G1B (Phosphatidylcholine 2-acylhydrolase 1B) concentration, immunoglobulin concentration and KRAS (Kirsten rat sarcoma viral oncogene) mutation load of collected pancreatic juice from different arms.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years old or older
* Diagnosis: CT, MRI, transabdominal ultrasound or other imaging examinations showed a pancreatic mass, and 3 endoscopists agreed on the diagnosis of suspected pancreatic cancer
* EUS-FNA is required to perform further treatment strategy
* The patient can understand the study protocol, is willing to participate in the study and can provide written informed consent

Exclusion Criteria:

* The patient's clinical and imaging features do not support the diagnosis of suspected pancreatic cancer, judged by 3 endoscopists
* The patient refuses to have EUS-FNA
* The patient is unsuitable for EUS-FNA because of his/her general condition, or contraindicated for anesthesia
* The patient's imaging suggests severe pancreatic duct obstruction
* The patient cannot understand the conditions and objectives of this study, or refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-12-30 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
KRAS mutation | The collected pancreatic juice will be tested in 6 months.
  Consistency of KRAS mutation detection results in genomic DNA of pancreatic tissue and cell-free DNA in pancreatic juice

SECONDARY OUTCOMES:
PLA2G1B concentration | The collected pancreatic juice will be tested in 6 months.
  PLA2G1B concentration of collected pancreatic juice of patients in different arms
Immunoglobulin (Ig) concentration | The collected pancreatic juice will be tested in 6 months.
  Immunoglobulin (Ig) concentration of collected pancreatic juice of patients in different arms
KRAS mutation load | The collected pancreatic juice will be tested in 6 months.
  KRAS mutation load detected of collected pancreatic juice of patients in different arms
cfDNA concentration | The collected pancreatic juice will be tested in 6 months.
  cfDNA concentration of pancreatic juice
DNA concentration of pancreatic juice | The collected pancreatic juice will be tested in 6 months.
  Genomic DNA concentration of exfoliated cells of pancreatic juice
Weight | The pancreatic juice will be weighed instantly 1 day (once) collected by EUS
  weight in grams of collected pancreatic juice of patients in different arms

CONTACTS AND LOCATIONS:
Overall Officials: Xi Wu, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No